CLINICAL TRIAL: NCT04525196
Title: Physical Activity in Dialysis: Clinical and Biological Impact
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dialyse
Record Dates: First submitted 2020-07-29; First posted 2020-08-25 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity. (Experimental): Patients will benefit a physical activity program during their dialysis session.
  Interventions: Other: Physical activity.
- No physical activity. (No Intervention): Patients will have access to their dialysis sessions without additional physical activity.

INTERVENTIONS:
Other: Physical activity. — The procedure under study (physical activity program) will include, each week for 12 months, two sessions dedicated to the development of aerobic capacity and a muscle building session.
  The experimental group will therefore be offered 3 sessions of Physical Activity (PA) per week. The PA will be positioned in the first two hours after the start of the dialysis session. Each session will include 5 minutes of general warm-up, then 15 minutes of PA itself and finally 5 minutes of cool down period. The PA time itself will be increased as the sessions progress, according to the progress and improvement of physical capabilities of patients.
  Arms: Physical activity.

SUMMARY:
Physical inactivity is known to increase the risk of developing many diseases as cardiovascular diseases, diabetes, some cancers, and other chronic diseases.

The impact of the inactivity is even higher in a fragile population as patients with Chronic Renal Failure (CRF) who need dialysis. This can lead to serious adverse events during the lifetime of these patients, such as arteriopathy which can result in amputation, deterioration of general condition, loss of independence and depression of wasting away.

Despite the need to promote physical activity in this population of hemodialysis patients with CRF, little is known about the effects of a supervised physical activity conducted in these patients.

With this study, the investigators propose to assess the effects of a physical activity program on several parameters, in hemodialysis subjects.

DETAILED DESCRIPTION:
The health risk of a sedentary and inactive lifestyle is known in the general population, increasing the risk of diabetes (+ 25%), obesity, arterial hypertension, stroke, myocardial infarction and the development of certain cancers.

Sedentary lifestyle therefore decreases longevity and life expectancy by 5 and 8 years respectively.

At the same time, the benefits of physical activity (PA) are recognized (the list is not exhaustive):

* Factor for improving physical capacity,
* Preventive effect on many cardiovascular risk factors,
* Improvement of psychological well-being (anxiety, depression, stress, etc.),
* Cognitive functions, reduction in the rate of certain cancers (colon and breast mainly),
* Reduction of oxidative stress. The High Authority of Health (HAS) recognizes physical activity as a therapy on its own in the prevention of chronic diseases after having noticed the harmful effects of physical inactivity (PI) on life expectancy.

PI is believed to be responsible for 1.9 million deaths worldwide each year, increasing public health costs, estimated at 150-300 euros per year and per citizen.

The population of patients with Chronic Renal Failure (CRF) on dialysis has a low physical capacity, a low level of PA decreasing as the number of years of dialysis increases.

These parameters are correlated with mortality: a critical number of steps of less than 4000 per day, or activity less than 50 minutes per day without dialysis significantly worsens mortality.

The association between mortality and level of PA is linear and this linearity is maintained over time.

CRF and dialysis promote catabolic factors in metabolism, decline in muscle mass and strength to sarcopenia (associated with inflammation, hypoandrogenism, intakes of inadequate protein, metabolic acidosis, insulin resistance and inactivity).

The decline in physical performance promotes falls, fractures, loss of autonomy, the number of hospitalizations which indirectly increases public health costs.

Several studies have shown the benefit of developing a per-dialytic PA program providing benefits in quality of life, physical capacity, reduction of hypotension blood pressure, depression, and VO2 max. Resistance exercise also improves muscle mass and strength.

PA acts as a cardioprotector by lowering total cholesterol, triglycerides, improving blood pressure profile, and consequently reducing the number of cardiovascular events on a follow-up of 2 years.

Finally, the DOPPS 2009-2011 observational study demonstrates the link between the level of physical aerobic activity and the parallel decline in mortality.

In addition, peripheral vascular and arterial complications are common in patients with CRF and dialysis. The prevalence of symptomatic Obstructive Arterial Disease of the Lower Limbs is estimated between 20% and 25% but it reaches 40% in the Japanese study of Matsuzawa, and 70% if associating the numerous asymptomatic patients.

Associated with the aging of the population and increasing sedentary lifestyle, we are faced with the appearance of extremely serious ischemic trophic disorders, difficult to treat, despite taking appropriate medical, surgical and cicatricial load often resulting in amputation, deterioration of general condition, loss of independence, depression of wasting away.

There is also an increased risk of associated cardiovascular mortality even in asymptomatic patients. The more severe the arterial disease is, greater the risk is. Thus, patients with critical ischemia have a one-year mortality of 25%.

Despite the importance of these data, associated with the individual consequences following amputations, the medical interest in this pathology is relatively low, and there are only few studies in hemodialysis subjects.

Exercise, especially walking, is recommended for patients at the stage of intermittent claudication. A meta-analysis performed in the general population showed that gait training improved walking ability by 150%.

The main objective of this study is to assess the clinical benefit of a physical activity program in terms of performance on the 6-minute walk test.

One of the secondary objectives of this study will be to assess the impact of a PA program on the occurrence of Obstructive Arterial Disease of the Lower Limbs. The investigators want to check whether the implementation of a program of per-dialytic physical activity would improve the microcirculation of the lower limbs and reduce the complications of arteritis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or over.
* Patient on hemodialysis.
* Patient in sufficient clinical condition allowing performing physical activity sessions during dialysis, according to the judgment of the investigator.
* Patient who was informed of the study and who gave his informed consent.
* Patient benefiting from a mandatory social security.

Exclusion Criteria:

* Recent myocardial infarction (<1 month).
* Rheumatological pathology which does not allow pedaling.
* Unmatched amputation of the lower limbs.
* Patients under legal protection.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2025-07-29 (Estimated); Study Completion 2025-07-29 (Estimated)

PRIMARY OUTCOMES:
The clinical impact of a physical activity program on the walking capacity. | Baseline.
  Measure and evolution of the performance to the 6 minutes walking test.
The clinical impact of a physical activity program on the walking capacity. | 6 months after the inclusion.
  Measure and evolution of the performance to the 6 minutes walking test.

SECONDARY OUTCOMES:
The clinical impact of a 12 month physical activity program on the aeroby capacity of the patients. | At the randomization visit, and 12 months after the inclusion.
  Measure and evolution of the performance to the 6 minutes walking test.
The clinical impact of a physical activity program on the muscle binding. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the extension force of the lower limbs.
The clinical impact of a physical activity program on the muscle binding. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the extension force of the handgrip.
The clinical impact of a physical activity program on the muscle binding. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the extension force of the elbow flexion.
The clinical impact of a physical activity program on the muscle binding. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the extension force of the sit/stand up test.
The impact of a physical activity program on the nutritional status. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the weight in kg.
The impact of a physical activity program on the nutritional status. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the BMI in kg/m².
The impact of a physical activity program on the nutritional status. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the body surface given in m².
The impact of a physical activity program on the nutritional status. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the active cell mass in kg.
The impact of a physical activity program on the nutritional status. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the muscle mass in kg.
The impact of a physical activity program on the nutritional status. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the mass index lean in kg.
The impact of a physical activity program on the nutritional status. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the albuminemia in g/L.
The impact of a physical activity program on the nutritional status. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the pre-albuminemia in g/L.
The impact of a physical activity program on the nutritional status. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the nPCR (Normalized Protein Catabolic Rate) in g/kg/day.
The impact of a physical activity program on the nutritional status. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the creatinine in mmol/L.
The impact of a physical activity program on the Obstructive Arterial Disease of the Lower Limbs. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the systolic pressure index and the systolic pressure of the toe measured by the SYSTOE, the number of revasularisations, the number of ischemic wounds, the number of amputations, and the number of deaths linked to the Obstructive Arterial Disease of the Lower Limbs.
To assess the impact on a physical activity program on the biological parameters. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the hemoglobin in g/dl.
The impact on a physical activity program on the biological parameters. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the CRP in μg/mL.
The impact on a physical activity program on the biological parameters. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Measure and evolution of the PTH in pg/mL.
To assess the impact of a physical activity program on the quality of life. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Evolution of the score obtained at the SF-36 questionnaire.
The impact of a physical activity program on the survival. | At the randomization visit, 6 months after the inclusion and 12 months after the inclusion.
  Evolution of the vital status.
To assess the impact of a physical activity program on the the relationship between caregivers and patients, the creation of social ties and "coping" (the ability to cope and adapt in response to stress) | At the randomization visit, and 6 months after the inclusion.
  Evolution of the score obtained at the WCC-R questionnaire.
The compliance with physical activity. | After each physical activity session performed by the patient.
  Development of aerobic capacity: the duration and, if applicable, the resistance level will be specified for each session.
The compliance with physical activity. | After each physical activity session performed by the patient.
  Muscle strengthening: the number of repetitions performed and the resistance level will be specified for each session.
The tolerance to physical activity. | 1 year, during each physical activity session.
  Adverse events: collection of the frequency and severity. Collection of the adverse events related to the PA program (group experimental only).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Bouchard, Marseille
  - Polyclinique les Fleurs, Ollioules

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pedersen BK. Muscles and their myokines. J Exp Biol. 2011 Jan 15;214(Pt 2):337-46. doi: 10.1242/jeb.048074. PMID 21177953
- [Background] Vina J, Sanchis-Gomar F, Martinez-Bello V, Gomez-Cabrera MC. Exercise acts as a drug; the pharmacological benefits of exercise. Br J Pharmacol. 2012 Sep;167(1):1-12. doi: 10.1111/j.1476-5381.2012.01970.x. PMID 22486393
- [Background] Sietsema KE, Amato A, Adler SG, Brass EP. Exercise capacity as a predictor of survival among ambulatory patients with end-stage renal disease. Kidney Int. 2004 Feb;65(2):719-24. doi: 10.1111/j.1523-1755.2004.00411.x. PMID 14717947
- [Background] Kopple JD, Kim JC, Shapiro BB, Zhang M, Li Y, Porszasz J, Bross R, Feroze U, Upreti R, Kalantar-Zadeh K. Factors affecting daily physical activity and physical performance in maintenance dialysis patients. J Ren Nutr. 2015 Mar;25(2):217-22. doi: 10.1053/j.jrn.2014.10.017. PMID 25701942
- [Background] Panaye M, Kolko-Labadens A, Lasseur C, Paillasseur JL, Guillodo MP, Levannier M, Teta D, Fouque D. Phenotypes influencing low physical activity in maintenance dialysis. J Ren Nutr. 2015 Jan;25(1):31-9. doi: 10.1053/j.jrn.2014.07.010. Epub 2014 Oct 8. PMID 25304464
- [Background] Matsuzawa R, Roshanravan B, Shimoda T, Mamorita N, Yoneki K, Harada M, Watanabe T, Yoshida A, Takeuchi Y, Matsunaga A. Physical Activity Dose for Hemodialysis Patients: Where to Begin? Results from a Prospective Cohort Study. J Ren Nutr. 2018 Jan;28(1):45-53. doi: 10.1053/j.jrn.2017.07.004. Epub 2017 Sep 8. PMID 28893466
- [Background] Matsuzawa R, Matsunaga A, Wang G, Kutsuna T, Ishii A, Abe Y, Takagi Y, Yoshida A, Takahira N. Habitual physical activity measured by accelerometer and survival in maintenance hemodialysis patients. Clin J Am Soc Nephrol. 2012 Dec;7(12):2010-6. doi: 10.2215/CJN.03660412. Epub 2012 Sep 13. PMID 22977216
- [Background] Johansen KL, Kaysen GA, Dalrymple LS, Grimes BA, Glidden DV, Anand S, Chertow GM. Association of physical activity with survival among ambulatory patients on dialysis: the Comprehensive Dialysis Study. Clin J Am Soc Nephrol. 2013 Feb;8(2):248-53. doi: 10.2215/CJN.08560812. Epub 2012 Nov 2. PMID 23124787
- [Background] Heiwe S, Jacobson SH. Exercise training in adults with CKD: a systematic review and meta-analysis. Am J Kidney Dis. 2014 Sep;64(3):383-93. doi: 10.1053/j.ajkd.2014.03.020. Epub 2014 Jun 7. PMID 24913219
- [Background] Manfredini F, Mallamaci F, D'Arrigo G, Baggetta R, Bolignano D, Torino C, Lamberti N, Bertoli S, Ciurlino D, Rocca-Rey L, Barilla A, Battaglia Y, Rapana RM, Zuccala A, Bonanno G, Fatuzzo P, Rapisarda F, Rastelli S, Fabrizi F, Messa P, De Paola L, Lombardi L, Cupisti A, Fuiano G, Lucisano G, Summaria C, Felisatti M, Pozzato E, Malagoni AM, Castellino P, Aucella F, Abd ElHafeez S, Provenzano PF, Tripepi G, Catizone L, Zoccali C. Exercise in Patients on Dialysis: A Multicenter, Randomized Clinical Trial. J Am Soc Nephrol. 2017 Apr;28(4):1259-1268. doi: 10.1681/ASN.2016030378. Epub 2016 Dec 1. PMID 27909047
- [Background] Olvera-Soto MG, Valdez-Ortiz R, Lopez Alvarenga JC, Espinosa-Cuevas Mde L. Effect of Resistance Exercises on the Indicators of Muscle Reserves and Handgrip Strength in Adult Patients on Hemodialysis. J Ren Nutr. 2016 Jan;26(1):53-60. doi: 10.1053/j.jrn.2015.06.006. Epub 2015 Aug 8. PMID 26264173
- [Background] Isnard-Rouchon M, Coutard C. [Exercise as a protective cardiovascular and metabolic factor in end stage renal disease patients]. Nephrol Ther. 2017 Dec;13(7):544-549. doi: 10.1016/j.nephro.2017.01.027. Epub 2017 Nov 7. French. PMID 29126841
- [Background] Lopes AA, Lantz B, Morgenstern H, Wang M, Bieber BA, Gillespie BW, Li Y, Painter P, Jacobson SH, Rayner HC, Mapes DL, Vanholder RC, Hasegawa T, Robinson BM, Pisoni RL. Associations of self-reported physical activity types and levels with quality of life, depression symptoms, and mortality in hemodialysis patients: the DOPPS. Clin J Am Soc Nephrol. 2014 Oct 7;9(10):1702-12. doi: 10.2215/CJN.12371213. Epub 2014 Oct 2. PMID 25278548
- [Background] Matsuzawa R, Aoyama N, Yoshida A. Clinical Characteristics of Patients on Hemodialysis With Peripheral Arterial Disease. Angiology. 2015 Nov;66(10):911-7. doi: 10.1177/0003319715572678. Epub 2015 Feb 18. PMID 25694516
- [Background] Gerhard-Herman MD, Gornik HL, Barrett C, Barshes NR, Corriere MA, Drachman DE, Fleisher LA, Fowkes FGR, Hamburg NM, Kinlay S, Lookstein R, Misra S, Mureebe L, Olin JW, Patel RAG, Regensteiner JG, Schanzer A, Shishehbor MH, Stewart KJ, Treat-Jacobson D, Walsh ME. 2016 AHA/ACC Guideline on the Management of Patients With Lower Extremity Peripheral Artery Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2017 Mar 21;69(11):1465-1508. doi: 10.1016/j.jacc.2016.11.008. Epub 2016 Nov 13. No abstract available. PMID 27851991